CLINICAL TRIAL: NCT06793878
Title: School-Based Living In Families With Emotions Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daphne Holt, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019P003154
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Living in Families With Emotions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental): Living in Families with Emotions (LIFE)
  Interventions: Behavioral: Living in Families With Emotions

INTERVENTIONS:
Behavioral: Living in Families With Emotions — This is an 8-week group-based psychosocial intervention teaching adolescents how to recognize their feelings, manage them, and talk about emotions through group discussions, live exercises, and games. The adolescents' caregivers are also provided with the same information, through two live sessions.

SUMMARY:
The overall purpose of this study is to identify adolescents who are at-risk for psychosis, as evidenced by endorsement of mild-to-moderate, sub-syndromal symptoms, and provide them with a potentially preventive intervention aimed at enhancing resilience.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adolescents from the Boston area who are in middle school at the time of enrollment;
2. Enrolled in a school where study screening is taking place;
3. Have a parent or legal guardian who is able and willing to provide written informed consent;
4. Competent and willing to provide written informed assent;
5. English language proficiency of parent/guardian and participant;
6. Response of "yes, definitely" or "maybe" to auditory hallucinations, visual hallucinations, or paranoia on the Adult Psychotic-like Symptom Checker (APSS);
7. Able to safely participate in the protocol and appropriate for outpatient level of care, in the opinion of the investigator.

Exclusion Criteria:

1. Current DSM-V diagnosis with serious active symptoms (such as active psychotic symptoms, current suicidality, serious active alcohol or substance use, marked deterioration in functioning over the prior month) that necessitates close monitoring or individual therapy and/or inpatient or partial hospitalization;
2. Current enrollment in psychological or behavioral health treatment;
3. Current use of psychotropic medications (other than stimulants) prescribed by a physician;
4. Severe developmental delays (including, but not limited to, Autism Spectrum Disorder, Intellectual Disability, and Down Syndrome).

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility and Acceptability | Before the intervention and 8 weeks later
  This measure includes participant (both adolescent and parent/caregiver) attendance, with more attendance of the intervention indicating better feasibility and acceptability.
Adolescent Psychotic-Like Symptom Screener (APSS) | Before the intervention, 8 weeks later, 6 months later, and 12 months later
  The APSS is a 7-item measure assessing the presence of: visual and auditory hallucinations, paranoia, grandiosity, delusions of control, mind reading, and delusions of reference. Items are scored on a 3-point Likert scale (0=No, never, 0.5=Maybe, or 1=Yes, definitely) and are then summed for a total score.

SECONDARY OUTCOMES:
The Center for Epidemiological Studies Depression scale for children (CES-DC) | Before the intervention, 8 weeks later, 6 months later, and 12 months later
  The CES-DC is a 20-item self-report measure rated on a 4-point Likert scale that captures symptoms of depression within the past week, with higher ratings representing more severe depression.
Concise Health Risk Tracking Self-Report (CHRT-SR) | Before the intervention, 8 weeks later, 6 months later, and 12 months later
  The CHRT-SR measures suicidal thoughts and behaviors using 14-items, with higher ratings indicating more suicidal thoughts and behaviors.
Screen for Child Anxiety Related Disorders (SCARED) | Before the intervention, 8 weeks later, 6 months later, and 12 months later
  The SCARED is a 41 item measure to capture anxiety. It is rated on a 3 point Likert scale (not true or hardly ever true, somewhat true or sometimes true, or very true or often true).
The Child Behavior Checklist (CBCL) | Before the intervention, 8 weeks later, 6 months later, and 12 months later
  Parents/caregivers rated the CBCL, a 113-item multiple choice self-report measure to capture psychiatric symptoms of the adolescent through parent/caregiver ratings.
The Penn Emotion Recognition Test (ER-40) | Before the intervention, 8 weeks later, 6 months later, and 12 months later
  This is a 15-minute computer-based task which involves identifying which emotion (neutral, sad, happy, angry, or scared) is being expressed in 40 (half male and half female presenting) online images of faces to measure facial emotion recognition.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States